CLINICAL TRIAL: NCT04234308
Title: Clinical, Mechanical, and Histological Properties of Absorbable and Nonabsorbable Suture Materials Used in Periodontal and Dental Implant Surgery.
Brief Title: Properties of Absorbable and Nonabsorbable Suture Material in Dental Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Científica del Sur (Other)
Collaborators: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 010-2019-PRO8
Record Dates: First submitted 2020-01-11; First posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Suture Adverse Reaction; Suture; Complications, Mechanical; Suture Failure During Surgical Operation; Suture Related Complication; Suture Rupture; Suture; Complications, Infection or Inflammation; Suture Line Infection
Keywords: dental suture; suture infection; Mechanical properties; absorbable sutures; non-absorbable sutures; histological properties
MeSH Terms: conditions — Infections; Inflammation | interventions — Polyglycolic Acid; Catgut; Polytetrafluoroethylene; Nylons

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Polyglycolic Acid Absorbable suture (Experimental): Periodontal and periimplant flaps closed with at least one suture with Polyglycolic Acid Absorbable suture, synthetic, 4-0. (TAGUM®).
  Interventions: Drug: Polyglycolic Acid
- Chromic Gut Absorbable suture (Experimental): Periodontal and periimplant flaps closed with at least one suture with Chromic Gut Absorbable suture, natural, 4-0. (TAGUM®)
  Interventions: Drug: Catgut
- ePTFE Non absorbable suture (Experimental): Periodontal and periimplant flaps closed with at least one suture with ePTFE Non absorbable suture, synthetic, 4-0. (TAGUM®)
  Interventions: Drug: Polytetrafluoroethylene
- Nylon Non absorbable sutures (Experimental): Periodontal and periimplant flaps closed with at least one suture with Nylon Non absorbable sutures, synthetic, 4-0. (TAGUM®)
  Interventions: Drug: Polyamide

INTERVENTIONS:
Drug: Polyglycolic Acid — Periodontal and periimplant flaps closed with at least one suture with Polyglycolic Acid Absorbable suture, synthetic, 4-0. (TAGUM®).
  Arms: Polyglycolic Acid Absorbable suture
Drug: Catgut — Periodontal and periimplant flaps closed with at least one suture with Chromic Gut Absorbable suture, natural, 4-0. (TAGUM®)
  Arms: Chromic Gut Absorbable suture
Drug: Polytetrafluoroethylene — Periodontal and periimplant flaps closed with at least one suture with expanded Polytetrafluoroethylene Non absorbable suture, synthetic, 4-0. (TAGUM®)
  Other Names: ePTFE
  Arms: ePTFE Non absorbable suture
Drug: Polyamide — Periodontal and periimplant flaps closed with at least one suture with Nylon Non absorbable sutures, synthetic, 4-0. (TAGUM®)
  Other Names: Nylon
  Arms: Nylon Non absorbable sutures

SUMMARY:
A suture is a biomedical device that is made of natural or synthetic materials. Sutures are used to close tissue surfaces until wounds heal and regain their ability to withstand normal stresses. Although different suture materials are available for various dental procedures, clinicians commonly neglect to select sutures based on their mechanical properties and capabilities. Instead, clinicians rely on their clinical experience to determine which suture material will suffice for wound closure and healing. To our knowledge, there have been no published studies detailing the results of mechanical testing on sutures after clinical application. The aim of this study is to clinically, histologically, and mechanically assess the four common sutures used in periodontal and dental surgery, with the hopes of providing clinicians with a guide that will allow them to choose sutures based on the clinical, histological, mechanical properties that best fit the stress and strain applied to the wound.

ELIGIBILITY:
Inclusion Criteria:

Subject must have read, understood and signed the informed consent form. Subject must require either open flap debridement surgery or implant placement (one to three consecutive teeth replacement) surgery.

Subjects must be males or females who are a minimum of 20 years of age. No history of periodontal or implant surgery at the investigational area site within the past 12 months.

Periodontal probing depths ≥5 mm interdentally at the implant site. Subjects that received single interrupted sutures for flap closure following surgical procedures.

Exclusion Criteria:

* Subject is part of a vulnerable population will be excluded. Female subjects who are pregnant or lactating, or who intend to become pregnant during the study period following entrance into the study.

Subjects with a systemic disease that would preclude periodontal surgery. Subjects who are smokers or chew tobacco. Subjects that received periodontal dressing on the surgical area. Subjects with the presence of acute infectious lesions in the areas intended for surgery.

Subjects with conditions or circumstances, in the opinion of the Investigator, which would prevent completion of study participation or interfere with analysis of study results.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
healing changes around each suture material | 1 week, 2 weeks 1 month and 3 months after surgery.
  To determinate the healing changes around each suture material using the Healing Index of Landry and colleagues (1988)
Tensile and mechanical properties of each suture material | following 1 week of clinical application.
  Evaluation of the tensile mechanical properties of each suture material using a Chatilloin TCD200 jig attachment, and tensile load will be applied to each suture at 0.05N/mm per min. Each suture will be stretched to failure and the maximum load will be recorded in Newtons (N).
Biofilm formation around each suture material | following 1 week of clinical application.
  To determinate the biofilm formation around each suture material using PCR

SECONDARY OUTCOMES:
complications including erythema, edema, hematoma, infection, wound dehiscence, keloid or scar tissue | 1 week, 2 weeks, 1 month and 3 months after surgery.
  To determinate the presence of complications including erythema, edema, hematoma, infection, wound dehiscence, keloid or scar tissue
plaque adherence over sutures, number of sutures present and number of stable (untied) sutures | 1 week after surgery.
  To determinate the plaque adherence over sutures, number of sutures present and number of stable (untied) sutures
  • Plaque adherence over sutures. This will be classified as following: 0: no debris or plaque present;
  1. soft debris or plaque covering not more than one third of the sutures,
  2. soft debris or plaque covering more than one third of the exposed suture;
  3. soft debris of plaque covering more than two thirds of the exposed sutures.
subject satisfaction | 1 week and 3 months following surgery.
  To determinate subject pain/satisfaction using a Visual Analogue Scale (VAS) at Visits 2 and 5. The VAS will be given to the subject in order to rate the satisfaction on a scale from 0 to 10, where 10 is the highest level of pain/satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ismael Khouly, PhD, Principal Investigator — New York University

IPD SHARING:
Plan to Share IPD: No